CLINICAL TRIAL: NCT05782361
Title: A Proof-of-concept Trial With Safety Run of Tepotinib and Pembrolizumab in NSCLC Patients With and Without MET Exon 14 Mutations (POTENT)
Brief Title: POTENT - Tepotinib in Combination With Pembrolizumab in NSCLC
Acronym: POTENT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR5558
Record Dates: First submitted 2023-01-13; First posted 2023-03-23 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer; Non Small Cell Lung Cancer
Keywords: tepotinib; pembrolizumab; lung cancer; MET inhibition; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — tepotinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A- Escalation (Experimental): The safety run-in part of the study will enrol 6-12 patients. Tepotinib will be given to patients daily for three weeks. After thee weeks, patients will be given pembrolizumab immunotherapy on a 21-day cycle along side tepotinib daily.
  Dose de-escalation of Tepotinib only will be performed in in Part A.. Should dose level 1 (500mg OD) be deemed non-tolerable by the SRC then a single dose de-escalation to dose level -1 (250mg OD) may be performed. Alternative dosing schedules may be explored. Recruitment into Part A will be staggered such that at least 7 days elapse between treatment of the 1st and 2nd patient of each dose level. In the dose confirmation phase, the study will first evaluate the dose level 1 with 3 patients, expanding to a maximum of 6 evaluable patients. If needed, a maximum of 6 patients will be evaluate in the dose level -1.
  Recruitment to this arm is closed.
  Interventions: Drug: Tepotinib; Drug: Pembrolizumab
- Part B- Expansion (Experimental): The expansion part of the study will enrol 13-26 patients with NSCLC and MET exon 14 skipping mutations. The combination of tepotinib and pembrolizumab will be tested throughout this part of the study. The first cycle will test the safety run-in of tepotinib followed by the introduction of combination with pembrolizumab from cycle 2 onwards.
  Recruitment to this arm is open.
  Interventions: Drug: Tepotinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Tepotinib — Tepotinib hydrochloride hydrate will be supplied as film coated tablets. The 250 mg oval, white-pink film-coated tablets contain the excipients mannitol, microcrystalline cellulose, crospovidone, magnesium stearate, colloidal silicon dioxide, and Opadry II pink. All formulations are intended for oral administration. Refer to pharmacy manual for formulation and strength information.
Drug: Pembrolizumab — Pembrolizumab Solution for Infusion 100 mg/vial is a liquid drug product supplied as a clear to opalescent solution, essentially free of visible particles, in Type I glass vials and manufactured using the fully formulated drug substance with L-histidine as buffering agent, polysorbate 80 as surfactant, and sucrose as stabilizer/tonicity modifier.
  Pembrolizumab Solution for Infusion can be further diluted with normal saline or 5% dextrose in the concentration range of 1 to 10 mg/mL in IV containers made of polyvinyl chloride (PVC) or non-PVC material.
  Other Names: MK-3475

SUMMARY:
This clinical study is looking at the combination of two experimental drugs called tepotinib and pembrolizumab. Pembrolizumab, also known as Keytruda, is licenced and available by prescription to treat a variety of cancers. Tepotinib is currently licensed in the UK for use in non-small cell lung cancer (NCSLC) and is being investigated for this purpose.

Cancer immunotherapy drugs hold great promise but still do not work for many patients. Laboratory studies on cancers that do not respond well to immunotherapy reveal that most of these tumours do not have any immune cells. This suggests that the cancer has successfully hidden itself and avoided being recognised by the immune system. This study aims to use a novel approach using a targeted drug, tepotinib, to target the gene involved with NSCLC.

Tepotinib is a type of drug called a kinase inhibitor. Kinase inhibitors are a newer type of drug being used to try to treat cancers. They act by blocking some of the chemical messengers that are part of the signalling process within cancer cells that control their growth. Tepotinib is used in adults to treat NSCLC that can have certain abnormal changes in the mesenchymal-epithelial transition factor gene (MET) and which has spread and/or cannot be removed by surgery. The changes in the MET gene can make an abnormal protein which can lead to uncontrolled cell growth and cancer. By blocking this abnormal protein, tepotinib may slow or stop the cancer from growing as well as potentially shrinking the cancer. This study will include patients with and without the MET exon 14 mutations.

In this clinical study, the investigators aim to test our ideas in a small number of people for the first time, specifically in those patients with cancers which do not respond to cancer immunotherapy.

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients aged 18 or over; 2. Non-small cell lung cancer histologically confirmed; 3.

Part A:

Either

a) Exon 14 MET mutation (on tissue or ctDNA testing); b) Patients have not received prior immunotherapy; c) Patients who have received previous MET inhibitor therapy must have PD-L1 TPS≥50% (not required in those naïve to MET inhibitors).

Or a) Patient has received at least one line of systemic anticancer therapy for metastatic disease; b) Patient has received at least two cycles of immune checkpoint inhibitor and has demonstrated disease progression within 12 weeks of last dose.

4.

Part B:

Cohort 1

a) Exon 14 MET mutation (on tissue or ctDNA testing); b) Patients have not received prior immunotherapy; c) Patients who have received previous MET inhibitor therapy must have PD-L1 TPS≥50% (not required in those naïve to MET inhibitors).

5. Measurable disease as assessed by iRECIST 6. Life expectancy of at least 12 weeks. 7. World Health Organisation (WHO) performance status of 0 or 1(Appendix 1). 8. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) prior to the patient's first dose of IMP.

Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x (ULN) unless raised due to tumour in which case up to 5 x ULN is permissible Renal function

Either:

Serum creatinine ≤ 1.5 x upper limit of normal (ULN); Or GFR ≥ 50 mL/min (uncorrected value) Calculated creatinine clearance (using the Wright, Cockcroft & Gault formula) Coagulation INR < 1.5 APTT <1.5x ULN Unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

9. Written (signed and dated) study informed consent and be capable of co-operating with treatment and follow-up. If patient does not comply with study procedures such that safety of the trial is affected then they will be withdrawn from the study.

10. Female patients with reproductive potential must have a negative urine or serum pregnancy test performed within 7-days prior to start of trial.

Exclusion Criteria:

1. Endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) and four weeks for investigational medicinal products), except for bisphosphonates or RANK ligand antagonists that are permitted for the management of bone metastases. Radiotherapy at radical doses within 6 months and at palliative doses within 2 weeks. Patients already receiving tepotinib prior to trial are not required to cease tepotinib prior to trial entry.

2. Ongoing Grade 2 or greater toxicities of previous treatments. Exceptions to this are alopecia and ongoing anticoagulation therapy due to prior thromboembolic episodes.

3. History of ILD or interstitial pneumonitis requiring steroid administration. 4. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom) for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible.

5. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using a barrier method of contraception [condom plus spermicide] or to sexual abstinence effective from the first administration of IMP throughout the trial and for six months afterwards. Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel or sexual abstinence). Men with pregnant or lactating partners must be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure of the foetus or neonate.

NB. Abstinence is only considered to be an acceptable method of contraception when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

6.

Known untreated or active central nervous system (CNS) metastases (progressing or requiring corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided they meet all of the following criteria:

* Evaluable or measurable disease outside the CNS is present.
* Radiographic stability upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the baseline disease assessment
* Not requiring corticosteroids. 7. Major surgery within four weeks of the first dose of study treatment. 8. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.

Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).

10. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment.

11. Has an active autoimmune disease that has required systemic treatment in past 3 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with a history of inflammatory bowel diseases such as Crohn's disease or ulcerative colitis will be excluded from the study. Patients with Sjogren's syndrome will not be excluded from the study. In addition, patients that experienced a Grade 2 or higher immune-related AEs on treatment with immunotherapy will be excluded from the study. Patients with inactive autoimmune disease which has previously required systemic therapy, may be considered on a case-by-case basis after discussion with the chief investigator.

12. Has a known history of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins.

13. Has received a live vaccine within 30 days of planned start of study therapy. Note: The killed virus vaccines used for seasonal influenza vaccines for injection are allowed; however intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.

14. Has experienced hypersensitivity to tepotinib, pembrolizumab or any of their excipients.

15.

Any of the following cardiac criteria:

* Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 consecutive electrocardiograms (ECGs) within 5 minutes of each other. Known congenital QT syndrome or history of torsades de pointes.
* Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG, e.g. complete left bundle branch block, third degree heart block. Controlled atrial fibrillation is allowed.
* Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, angina pectoris, congestive heart failure New York Heart Association [NYHA Grade 2 or above], severe valvular disease, uncontrolled hypertension despite optimal therapy.

Prior bone marrow transplant or have had extensive radiotherapy to greater than 25% of bone marrow within eight weeks.

17. Current malignancies of other types, with the exception of adequately treated cone biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. An exception to this criteria are cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for three years or more and are deemed at negligible risk for recurrence, are eligible for the trial.

18. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase I study. Participation in an observational trial would be acceptable.

19. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

20. Symptoms of active COVID-19 and/or documented active COVID-19 infection at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2028-03-08 (Estimated); Study Completion 2029-01-09 (Estimated)

PRIMARY OUTCOMES:
Anti-tumour activity evaluation (in Part B) | 24 Months
  Assessing the antitumour activity of tepotinib in combination with pembrolizumab using the overall response rate as defined by disease response using iRECIST

SECONDARY OUTCOMES:
Determination of MTD and RP2D | 12 Months
  Establishing the recommended Phase II dose (RP2D) of tepotinib in combination with pembrolizumab by determining a dose at which no more than one patient out of six patients at the same dose level experience a drug-related dose limiting toxicity (DLT).
Safety and tolerability of the combination of tepotinib with pembrolizumab | 24 Months
  Determining causality of each adverse event to the combination of tepotinib with pembrolizumab and grading severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
  Discontinuation rate defined as number of patients discontinuing IMP due to toxicity
Further anti-tumour activity evaluation | 24 Months
  Evaluating the further measures of antitumour activity of tepotinib in combination with pembrolizumab. Clinical benefit rate defined as the percentage of patient who have achieved complete response, partial response or stable disease according to iRECIST
Pharmacokinetics of Tepotinib investigating maximum plasma concentration | 12 Months
  Determination of the plasma levels of Tepotinib in Part A of the study, using validated assays
Pharmacodynamics investigating the change in markers of target inhibition | 36 Months
  Characterising the pharmacodynamics (PD) profile of tepotinib in combination with pembrolizumab. Determination of changes in markers of target inhibition and immune microenvironment in tumour and blood including T-cell subsets and PD-L1. Analysis will be conducted using the fluorescence activated cell sorting and multi-coloured immunofluorescence.
Pharmacodynamics investigating the change in ctDNA | 36 Months
  Characterising the change in circulating tumour DNA sequencing over trial period for emerging mechanisms of resistance. Determination of allele frequency of genomic aberrations including but not limited to MET, EGFR, BRAF and KRAS in plasma. ctDNA samples will be taken on Day 1 of every cycle.
Overall survival | 24 Months
  Progression-free survival defined as time from cycle 1 day 1 (C1D1) to progressive disease according to iRECIST or death from any cause. The progression-free survival time of patients still alive and progression-free will be censored on the date of their last RECIST assessment.
  Overall survival defined as time from C1D1 to death from any cause. Survival time of living patients will be censored on the last date of patient is known to be alive or lost to follow up. Overall survival defined as time from C1D1 to death from any cause. Survival time of living patients will be censored on the last date of patient is known to be alive or lost to follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Minchom, MD, Principal Investigator — Royal Marsden Hospital NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - DDU, Royal Marsden Hospital NHS Foundation Trust, Sutton, Surrey
  - University College London Hospitals NHS Foundation Trust, London
  - Lung Unit, Royal Marsden Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No